CLINICAL TRIAL: NCT02917018
Title: Effect of Different Doses of Dexmedetomidine on Stress Response and Emergence Agitation After Laparoscopic Cholecystectomy in Adults
Brief Title: Effect of Dexmedetomidine on Stress Response and Emergence Agitation During Laparoscopic Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MOHAMED F. MOSTAFA, lecturer of anesthesia and intensive care, faculty of medicine, Assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dexmed EA
Record Dates: First submitted 2016-09-05; First posted 2016-09-28 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Stress Response
Keywords: Dexmedetomidine; Stress response; Emergence agitation
MeSH Terms: conditions — Fractures, Stress; Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dexmedetomidine 1 (Active Comparator): patients will receive dexmedetomidine 1 mic/kg
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.75 (Active Comparator): patients will receive dexmedetomidine 0.75 mic/kg
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.5 (Active Comparator): patients will receive dexmedetomidine 0.5 mic/kg
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Group I will receive 1 ug/kg, group II will receive 0.75 ug/kg and group III will receive 0.5 ug/kg) diluted to 50 ml NaCl 0.9% by syringe pump over 20 minutes before end of surgery.

SUMMARY:
Emergence agitation is a post-anesthetic phenomenon that develops in the early phase of general anesthesia recovery, and is characterized by agitation, confusion, disorientation, and possible violent behavior. The incidence of emergence agitation is less common in adults as compared to pediatric patients. It may lead to serious consequences for the patient such as bleeding, falling, removal of catheters and self extubation, which lead to further complications like hypoxia and aspiration.

Despite its common occurrence, unclear etiology, and serious sequelae, emergence agitation has rarely been studied in adults.

The stress response to surgery is an unconscious response to tissue injury. Activation of the sympathetic nervous system, increase of catabolic hormone release and pituitary gland suppression are considered a response to surgical stress, in clinical practice these activities cause changes in heart rate, blood pressure and biochemical fluctuations of noradrenaline, adrenaline, dopamine, and cortisol. Above all, these fluctuations prolong hospitalization and delay patients discharge.

Dexmedetomidine is a highly selective alpha-2 receptor agonist having sedative, analgesic and sympatholytic properties. Decreased stress response to surgery ensuring a stable hemodynamic state is a beneficial property of the agent. Peri-operative use of dexmedetomidine also decreases postoperative opioid consumption, pain intensity, and antiemetic therapy. However, the data related to the effects of dexmedetomidine on reducing agitation from general anesthesia in adults are limited.

DETAILED DESCRIPTION:
With no premedication, all patients will have pre-oxygenation for 3-5 minutes and intravenous access will be secured. NaCl 0.9% 4 ml/kg/h will be infused intraoperatively. General anesthesia will be induced by fentanyl 1 ug/kg, propofol 2 mg/kg and nimbex (cisatracurium) 0.15 mg/kg. Endotracheal intubation then will be done using oral ETT of appropriate size under direct laryngoscopy and secured at the angle of the mouth. Sevoflurane inhalational anesthetic (2-4 %) and nimbex 0.03 mg/kg will be used for maintenance of anesthesia. The lungs will be mechanically ventilated to keep intra-operative EtCo2 between 35-40 mmHg.

Intraoperative monitoring:

Routine monitors including ECG, non-invasive blood pressure, pulse oxymetry and EtCo2 will be recorded every 5 minutes during the intra-operative 20 minutes of the study drug administration. Bradycadia (heart rate ˂ 60 beat/minute) will be treated with iv atropine 0.5 mg. Hypotension (mean arterial blood pressure ˂ 60 mmHg) will be treated with iv ephedrine 5 mg increments. Duration of anesthesia, sevoflurane % and duration of surgery will be recorded.

At the end of surgery and stoppage of sevoflurane inhalation, neostigmine 0.04 mg/kg and atropine 0.02 mg/kg will be used for muscle relaxant reversal (Time 0 in the emergence process), patients will be extubated and transferred to the PACU for recovery and monitoring.

Assessment in PACU:

Routine monitoring will be continued during staying in PACU. During emergence, the level of agitation will be evaluated using the Ricker sedation-agitation scale (RSAS). The maximum level of agitation will be recorded for each patient at time 0, 5, 10, 20, 30, 60 and 120 minutes. Emergence agitation was defined as any score on the sedation-agitation scale ≥ 5. Dangerous agitation was defined as a sedation-agitation scale score = 7 (3). If dangerous agitation occurs, it will be treated with fentanyl 1 ug/kg.

Duration of stay in PACU will be recorded. Criteria for discharge from PACU will be applied according to the modified Aldrete scoring system. A score ≥ 9 was required for discharge.

Postoperative Analgesia:

The 10 points Visual Analogue Scale (VAS) for pain measurement will be used to assess the severity of postoperative pain. Score 0 indicates no pain and score 10 indicates severe pain. If VAS ≥ 4, rescue analgesia will be indicated. Perfalgan infusion will be used as supplemental analgesia. The first dose and the total amount in 24 hours of perfalgan will be recorded. Patient's satisfaction will be recorded at the end of the first 24 hours postoperatively.

Blood Sampling:

Venous blood samples will be collected from peripheral extremities away from the intravenous infused limb. Samples will be withdrawn 30 minutes pre-operatively, 30 minutes after skin incision, 2 and 24 hours after end of surgery. The blood samples will be centrifuged at 3500 ×g for at least 10 minutes and then serum samples will be eluted. Blood glucose level will be also recorded at the same times.

Statistical Analysis:

Statistical analysis will be conducted with SPSS version 20 (SPSS Inc., Chicago, IL, USA) for Windows. The results will be expressed as mean ± SD, range, percentage. P-values < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II Laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* Patients with cardiac disease, diabetes. reactive upper airway disease. allergies to dexmedetomidine. cognitive disorders. renal insufficiency. hepatic dysfunction. Chronic use of analgesics, cortisone or drugs known to interact with dexmedetomidine.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
serum cortisol level | 2 hours postoperative
  serum cortisol level will be measured at 2 hours postoperative

SECONDARY OUTCOMES:
post anesthetic emergence agitation | 2 hours postoperative
  RSAS score will be measured 2 hours postoperative
visual analogue score | 24 hours postoperative
  perfalgan will be given when visual analogue score ≥ 4

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Yossef, MD, Study Chair — assiut university, faculty of medicine
Locations (1):
- Assiut university hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided